CLINICAL TRIAL: NCT04475276
Title: Effect of Alpha Lipoic Acid on Non-alcoholic Fatty Liver Diseases: A Randomized Placebo-controlled Clinical Trial
Brief Title: Effect of Alpha Lipoic Acid on Non-alcoholic Fatty Liver Diseases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: All India Institute of Medical Sciences, Bhubaneswar (Other)
Responsible Party: Principal Investigator, Dr. Monalisa Jena, M.D., Associate Professor, All India Institute of Medical Sciences, Bhubaneswar
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: T/IM-F/19-20/16
Record Dates: First submitted 2020-07-10; First posted 2020-07-17 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: Non alcoholic fatty liver; Alphalipoic acid; Nutraceutic; Insulin resistance; Cytokeratin 18; Life style modification; Vitamin E
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: A randomized, parallel design placebo-controlled clinical trial
Who Masked: Participant, Care Provider
Masking Description: The patients and the physician will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Life style modification with the placebo will be given for 12 weeks
  Interventions: Drug: Placebo
- Alphalipoic acid (Experimental): Life style modification with Alpha lipoic acid in a dose of 600mg twice daily will be prescribed orally for 12 weeks
  Interventions: Drug: Alphalipoic acid

INTERVENTIONS:
Drug: Placebo — Lifestyle modification with placebo for 12 weeks
  Arms: Placebo
Drug: Alphalipoic acid — Lifestyle modification with Alphalipoic acid for 12 weeks
  Arms: Alphalipoic acid

SUMMARY:
In developed counties Non-alcoholic fatty liver disease (NAFLD) becomes the most common cause of chronic liver disease , but its prevalence in developing countries like India is also increasing (10 -20%).Till date, there is no US-FDA approved therapy for NAFLD but drugs like metformin, pioglitazone, sitagliptin, vildagliptin Vitamin E, silymarin, statins and ezetimibe have been studied along with life style modification. Life style modifications is the current modality of treatment of NAFLD. All the above-mentioned drugs have some beneficial effects with limited use due to its adverse effects in patients of NAFLD and the study results are non-conclusive. In this scenario, a safe hepatoprotective drug to be evaluated in NAFLD.Alpha-lipoic acid (ALA) or 6,8-thioctic acid, is an endogenous molecule which functions as an important co-factor for various enzyme complexes in mitochondria and plays an important role in energy metabolism. ALA is a nutraceutical agent which also has hepatoprotective and anti-inﬂammatory effects.ALA is a nutraceutic having anti-inflammatory and antioxidant effects and also increasing insulin sensitivity with lesser adverse effects. The relative scarcity of a promising therapy and non-conclusiveness of the previous studies open up an arena of further research using a nutraceutic in non-diabetic NAFLD. So, the present study is designed to evaluate safety and efficacy of ALA in non-diabetic NAFLD patients.

DETAILED DESCRIPTION:
In developed counties Non-alcoholic fatty liver disease (NAFLD) becomes the most common cause of chronic liver disease , but its prevalence in developing countries like India is also increasing (10 -20%). Most of the patients are diagnosed clinically and by increased serum transaminase and fatty changes in liver on abdominal ultrasound. Till date, there is no US-FDA approved therapy for NAFLD but drugs like metformin, pioglitazone, sitagliptin, vildagliptin Vitamin E, silymarin, statins and ezetimibe have been studied along with life style modification. Life style modifications is the current modality of treatment of NAFLD. All the above-mentioned drugs have some beneficial effects with limited use due to its adverse effects in patients of NAFLD and the study results are non-conclusive. In this scenario, a safe hepatoprotective drug to be evaluated in NAFLD.

Alpha-lipoic acid (ALA) or 6,8-thioctic acid, is an endogenous molecule which functions as an important co-factor for various enzyme complexes in mitochondria and plays an important role in energy metabolism. ALA is a nutraceutical agent which also has hepatoprotective and anti-inﬂammatory effects. Previous animal studies proved the hepatoprotective effect of alpha lipoic acid on various animal models. Inflammatory liver injury involves the production of inflammatory mediators like nitric oxide and TNF-alpha. Alpha -Lipoic acid significantly inhibits production of nitric oxide and TNF-alpha. The reduced production of nitric oxide and TNF-alpha in Kupffer cells may be involved in the hepatoprotective action conveyed by alpha-lipoic acid.It has been proved that ALA has potent anti - inflammatory and anti- oxidant properties.

Insulin resistance is associated with impaired hepatic cell damage, intrahepatic cholestasis, atherogenic dyslipidaemia and fibrosis in patients of NAFLD. Daily treatment with ALA for 28 days significantly improved insulin sensitivity performance in mice by decreasing insulin resistance, IL-6 levels, acetylcholinesterase enzyme activity and oxidative stress in liver. Various studies have shown that the ALA can efficiently improve insulin sensitivity and reverse the insulin resistance. Cytokeratin 18 (CK 18) is released into circulation as a consequence of oxidative stress, hepatocyte apoptosis or inflammation in response to lipid metabolism in NAFLD. CK - 18 level is higher in insulin resistance.

ALA is a nutraceutic having anti-inflammatory and antioxidant effects and also increasing insulin sensitivity with lesser adverse effects. The relative scarcity of a promising therapy and non-conclusiveness of the previous studies open up an arena of further research using a nutraceutic in non-diabetic NAFLD. So, the present study is designed to evaluate safety and efficacy of ALA in non-diabetic NAFLD patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed to have fatty liver grading 1, 2, 3 on abdominal ultrasound, mild to moderate elevation (<5 times elevated upper limit) of serum aminotransferase level.
* Patients aged 18-65 years of either sex.
* Treatment naïve patients or patients who had not taken any treatment for at least 4 weeks before inclusion

Exclusion Criteria:

* History of diabetes mellitus, decompensated liver disease, ascites, oesophageal varices.
* Drug abusers and Alcoholics.
* HBs Ag positive, Anti HCV and HIV, hereditary defects of iron, copper and alpha- 1 antitrypsin deficient patients.
* Hypothyroidism, obstructive sleep apnoea, total parenteral nutrition, short bowel syndrome, pancreatoduodenal resection which are secondary causes of NAFLD.
* Drug users such as corticosteroids, antiviral (nucleoside analogue), tetracycline, methotrexate, tamoxifen and amiodarone.
* Patients who are taking any antihyperlipidemic and anti-diabetic agents.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-02-23 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Abdominal ultrasound | 12 weeks
  the change in fatty liver grading in NAFLD assessed by abdominal ultrasound

SECONDARY OUTCOMES:
Insulin resistance | 12 weeks
  changes in insulin resistance by using HOMA IR after therapy
Lipid profile | 12 weeks
  Change in lipid profile (Total Cholesterol, HDL, LDL,Triglycerides, VLDL) after therapy
  •
Levels of glutathione reductase | 12 weeks
  changes in levels of glutathione reductase after therapy
levels of Cytokeratin-18 | 12 weeks
  changes in levels of Cytokeratin-18 after therapy
Levels of Alanine transaminase (ALT) | 12 weeks
  changes in Alanine transaminase units per litre after therapy
Levels of Aspartate transaminase (AST) | 12 weeks
  changes in Aspartate transaminase (AST)units per litre after therapy
Levels of Alkaline phosphatase (ALP) | 12 weeks
  changes in Alkaline phosphatase (ALP) in IU after therapy
Levels of Albumin and total protein. | 12 weeks
  changes in Albumin and total protein in gm/L after therapy
Levels of Bilirubin | 12 weeks
  changes in Bilirubin in μmol/L after therapy
Levels of total protein | 12 weeks
  changes in total protein in gm/L after therapy
Levels of Gamma-glutamyltransferase (GGT). | 12 weeks
  changes in Gamma-glutamyltransferase (GGT) units per liter after therapy
Levels of L-lactate dehydrogenase (LDH). | 12 weeks
  changes in L-lactate dehydrogenase (LDH) units per liter after therapy

CONTACTS AND LOCATIONS:
Overall Officials: Rituparna Maiti, MD, Study Director — Additional Professor
Locations (1):
- AIIMS, Bhubaneswar, Odisha, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hussain M, Majeed Babar MZ, Hussain MS, Akhtar L. Vildagliptin ameliorates biochemical, metabolic and fatty changes associated with non alcoholic fatty liver disease. Pak J Med Sci. 2016 Nov-Dec;32(6):1396-1401. doi: 10.12669/pjms.326.11133. PMID 28083033
- [Background] Patel SS, Siddiqui MS. Current and Emerging Therapies for Non-alcoholic Fatty Liver Disease. Drugs. 2019 Jan;79(1):75-84. doi: 10.1007/s40265-018-1040-1. PMID 30588564
- [Background] Cavestro C, Bedogni G, Molinari F, Mandrino S, Rota E, Frigeri MC. Alpha-Lipoic Acid Shows Promise to Improve Migraine in Patients with Insulin Resistance: A 6-Month Exploratory Study. J Med Food. 2018 Mar;21(3):269-273. doi: 10.1089/jmf.2017.0068. Epub 2017 Oct 4. PMID 28976801
- [Background] Fayez AM, Zakaria S, Moustafa D. Alpha lipoic acid exerts antioxidant effect via Nrf2/HO-1 pathway activation and suppresses hepatic stellate cells activation induced by methotrexate in rats. Biomed Pharmacother. 2018 Sep;105:428-433. doi: 10.1016/j.biopha.2018.05.145. Epub 2018 Jun 5. PMID 29879626
- [Background] Sadek KM, Saleh EA, Nasr SM. Molecular hepatoprotective effects of lipoic acid against carbon tetrachloride-induced liver fibrosis in rats: Hepatoprotection at molecular level. Hum Exp Toxicol. 2018 Feb;37(2):142-154. doi: 10.1177/0960327117693066. Epub 2017 Feb 21. PMID 29233029
- [Background] Singh SP, Misra B, Kar SK, Panigrahi MK, Misra D, Bhuyan P, Pattnaik K, Meher C, Agrawal O, Rout N, Swain M. Nonalcoholic fatty liver disease (NAFLD) without insulin resistance: Is it different? Clin Res Hepatol Gastroenterol. 2015 Sep;39(4):482-8. doi: 10.1016/j.clinre.2014.08.014. Epub 2014 Dec 17. PMID 25543522
- [Background] Ahuja S, Uniyal A, Akhtar A, Sah SP. Alpha lipoic acid and metformin alleviates experimentally induced insulin resistance and cognitive deficit by modulation of TLR2 signalling. Pharmacol Rep. 2019 Aug;71(4):614-623. doi: 10.1016/j.pharep.2019.02.016. Epub 2019 Feb 23. PMID 31176103
- [Background] He L, Deng L, Zhang Q, Guo J, Zhou J, Song W, Yuan F. Diagnostic Value of CK-18, FGF-21, and Related Biomarker Panel in Nonalcoholic Fatty Liver Disease: A Systematic Review and Meta-Analysis. Biomed Res Int. 2017;2017:9729107. doi: 10.1155/2017/9729107. Epub 2017 Feb 23. PMID 28326329
- [Background] Tomic D, Kemp WW, Roberts SK. Nonalcoholic fatty liver disease: current concepts, epidemiology and management strategies. Eur J Gastroenterol Hepatol. 2018 Oct;30(10):1103-1115. doi: 10.1097/MEG.0000000000001235. PMID 30113367
- [Background] Wu G, Li H, Fang Q, Zhang J, Zhang M, Zhang L, Wu L, Hou X, Lu J, Bao Y, Jia W. Complementary Role of Fibroblast Growth Factor 21 and Cytokeratin 18 in Monitoring the Different Stages of Nonalcoholic Fatty Liver Disease. Sci Rep. 2017 Jul 11;7(1):5095. doi: 10.1038/s41598-017-05257-5. PMID 28698650
- [Background] Schurks M, Glynn RJ, Rist PM, Tzourio C, Kurth T. Effects of vitamin E on stroke subtypes: meta-analysis of randomised controlled trials. BMJ. 2010 Nov 4;341:c5702. doi: 10.1136/bmj.c5702. PMID 21051774
- [Background] Dulai PS, Singh S, Patel J, Soni M, Prokop LJ, Younossi Z, Sebastiani G, Ekstedt M, Hagstrom H, Nasr P, Stal P, Wong VW, Kechagias S, Hultcrantz R, Loomba R. Increased risk of mortality by fibrosis stage in nonalcoholic fatty liver disease: Systematic review and meta-analysis. Hepatology. 2017 May;65(5):1557-1565. doi: 10.1002/hep.29085. Epub 2017 Mar 31. PMID 28130788
- [Background] Khalaf AA, Zaki AR, Galal MK, Ogaly HA, Ibrahim MA, Hassan A. The potential protective effect of alpha-lipoic acid against nanocopper particle-induced hepatotoxicity in male rats. Hum Exp Toxicol. 2017 Sep;36(9):881-891. doi: 10.1177/0960327116674526. Epub 2016 Nov 12. PMID 27827802
- [Background] Abdel-Daim MM, Taha R, Ghazy EW, El-Sayed YS. Synergistic ameliorative effects of sesame oil and alpha-lipoic acid against subacute diazinon toxicity in rats: hematological, biochemical, and antioxidant studies. Can J Physiol Pharmacol. 2016 Jan;94(1):81-8. doi: 10.1139/cjpp-2015-0131. Epub 2015 Jul 19. PMID 26550680